CLINICAL TRIAL: NCT02651545
Title: Teriflunomide (Aubagio) Effects on Cognitive and Vocational Outcomes, as Related to Neurodegeneration in Multiple Sclerosis: A Prospective, Observational, Single-blinded Study.
Brief Title: Effects of Teriflunomide (Aubagio) on Cognitive and Vocational Outcomes in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ralph H.B. Benedict, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 1116240
Record Dates: First submitted 2014-05-14; First posted 2016-01-11 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Relapsing MS patients: Thirty (30) relapsing MS patients new to teriflunomide therapy will be enrolled.
- Healthy Controls: A sample of 30 healthy control volunteers, matched on demographics with the treated group will be enrolled.

SUMMARY:
Cognitive impairment is common in MS and has devastating impact on functional activities. There is a great demand for medications that will enhance cognitive capacity in MS patients. The effect of teriflunomide on cognition and vocational capacity is unknown. The investigators will address these questions in a sample of 30 relapsing MS patients treated with teriflunomide. Cognitive impairment will be measured by calculating an information processing speed index and a memory composite index from conventional, validated neuropsychological tests as recommended by consensus opinion publications. Vocational performance will be monitored using a newly developed online survey called the Multiple Sclerosis Vocational Monitoring Survey (MSVMS). This study will elucidate the effect of teriflunomide on these important outcomes.

DETAILED DESCRIPTION:
Summary:

Objectives: The primary aim of this study is to define the effect of teriflunomide (Aubagio®) on cognitive abilities in patients with relapsing multiple sclerosis (MS). There are two secondary objectives, to [a] relate changes in cognition to vocational problems, and [b] determine MRI correlates of change in cognition, more specifically gray-matter (GM) volume metrics which the investigators believe reflect neurodegeneration.

Design: This is a prospective, observational, single-blinded, longitudinal study of teriflunomide effects on cognitive performance in MS patients over 24 months. Neuropsychological status and 3T (3 Tesla) MRI will be assessed at baseline, 12 months and 24 months. Vocational status will be assessed every three months via the internet. Statistical analysis will emphasize within-subjects changes in all metrics to maximize statistical power.

Study Population: Thirty (30) relapsing MS patients and 30 healthy controls (HC) will be enrolled in the study.

Outcomes: An information processing speed index and a memory composite index will be calculated from conventional, validated neuropsychological tests as recommended by consensus opinion publications. Conventional clinical metrics for overall neurological disability will also be assessed. Vocational performance will be monitored using a newly developed online survey called the Multiple Sclerosis Vocational Monitoring Survey (MSVMS). Regional GM atrophy, as defined by measurement of thalamic and cortical atrophy, will serve as neurodegeneration outcomes.

Significance of the research: The effect of teriflunomide on the development of cognitive impairment and vocational capacity is unknown. This study will elucidate the effect of teriflunomide on these important outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with MS according to McDonald criteria
* Age 18-60
* Have a relapsing disease course
* Have Expanded Disability Status Scale scores of 0-6.5
* Have a disease duration <20 years
* Treatment naïve to teriflunomide
* Be willing and able to comply with the study procedures for the duration of the trial
* Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study-related activities are carried out
* Normal kidney functioning (creatinine clearance >59)
* None of the exclusion criteria

Exclusion Criteria:

* MS patients with hepatic impairment
* Nursing mothers or pregnant women who will need to undergo 12 months follow-up
* Women of childbearing potential not using reliable contraception
* Patients currently treated with teriflunomide
* A clinically significant infectious or neurological (for Healthy Controls only) illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to treatment assignment
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol
* History of neurological disorder other than MS
* History of developmental learning disorder or other developmental anomaly
* History of major depressive disorder, or other psychiatric disorder that could impact cognitive capacity, preceding diagnosis of MS
* Current major depressive episode
* Other pathology related to MRI abnormalities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of 30 relapsing MS patients new to teriflunomide therapy will be enrolled. A sample 30 healthy control volunteers, matched on demographics with the treated group will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph HB Benedict, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Buffalo General Hospital, D3, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relapsing MS Patients | Healthy Controls
Started | 30 | 30
Completed | 7 | 17
Not Completed | 23 | 13

BASELINE CHARACTERISTICS:
Groups:
- MS Group: Multiple Sclerosis Patients Prescribed Aubagio
- Healthy Control Group: Healthy controls matched to the MS group
- Total: Total of all reporting groups
Arm/Group | MS Group | Healthy Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.53 (8.97) | 47.77 (11.27) | 48.65 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 5 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23 | 27 | 50
  African American | 7 | 1 | 8
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Symbol Digit Modalities Test Total correct [Mean (Standard Deviation); unit: score on a scale] — The Symbol Digit Modalities Test (SDMT) is a measure to assess cognitive processing speed. The SDMT presents a series of 9 symbols, each paired to a single digit in a key at the top of a stimulus page. Subjects say the number associated with each symbol as rapidly as possible. The examiner records the responses. The task continues for 90 seconds with staff recording responses. The total number of correct responses is known as "Total Correct" and is used as the unit of measure. Score may range from 0 correct (slow processing speed) to 110 correct (faster processing speed).
  score on a scale | 49.7 (10.6) | 58.9 (8.5) | 54.3 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Scale Score (EDSS)
Description: The Expanded Disability Status Scale (EDSS). 0-10 scale with higher scores indicating more severe disability.
Time Frame: 0, 12, and 24 months
Measure: Median (Inter-Quartile Range); unit: EDSS Score
Arm/Group | Relapsing MS Patients
Number analyzed (Participants) | 30
EDSS Score
  EDSS Score Month 0 | 3.0 [2.0 to 4.63]
  EDSS Score Month 12 | 3.0 [2.0 to 4.88]
  EDSS Score Month 24 | 2.5 [2.0 to 6.0]

2. Primary Outcome: Timed 25-foot Walk.
Description: Time it takes in seconds for patient to walk 25 feet. Higher times indicate slower ambulation.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
Seconds
  Month 0 | 7.3 (3.7) | 4.6 (0.8)
  Month 12 | 7.4 (3.1) | 4.9 (1.2)
  Month 24 | 6.9 (2.6) | 5.3 (1.0)

3. Primary Outcome: Nine-hole Peg Test
Description: The Nine-Hole Peg test is a measure of manual dexterity, where the time in seconds that it takes for patient to fill pegboard holes with pegs and remove them is recorded. Longer times indicate slower motor ability. The range in seconds to complete the nine-hole peg test ranges from 0-seconds to the ceiling value of 300 seconds.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
Seconds
  Month 0 | 25.1 (6.6) | 20.0 (2.2)
  Month 12 | 26.7 (7.5) | 19.3 (2.3)
  Month 24 | 26.8 (6.9) | 20.1 (2.7)

4. Primary Outcome: California Verbal Learning Test 2nd Edition Total Learning Score
Description: A measure of verbal learning and memory. Patient is read a list of 16 words 5 times and asked to recall the list each time. Score 0-80 with higher scores indicating better performance.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
score on a scale
  Month 0 | 50.5 (12.5) | 55.3 (9.7)
  Month 12 | 47.8 (16.5) | 54.2 (8.5)
  Month 24 | 49.1 (14.6) | 53.1 (7.7)

5. Primary Outcome: Brief Visuospatial Memory Test Revised Total Learning Score
Description: A measure of visual-spatial learning and memory. Patient is shown a display 3 times and asked to recall figures from the display. Score 0-36 with higher scores indicating better performance.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
score on a scale
  Month 0 | 20.0 (6.5) | 24.4 (6.3)
  Month 12 | 19.0 (7.1) | 23.7 (7.6)
  Month 24 | 20.0 (9.3) | 24.9 (5.9)

6. Primary Outcome: Symbol Digit Modalities Test Total Correct
Description: A measure of cognitive processing speed. Patient is shown a key with symbol-digit pairings and several rows of symbols with empty boxes beneath them. Patient is asked to respond with the numbers that are paired with each of the symbols as quickly and accurately as they can. Score 0-120 with higher scores indicating better performance.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
score on a scale
  Month 0 | 49.7 (10.6) | 58.9 (8.5)
  Month 12 | 47.3 (12.8) | 57.1 (11.6)
  Month 24 | 48.9 (10.1) | 59.6 (11.0)

7. Secondary Outcome: Change in Vocational Status
Description: Vocational Status assessed by the Buffalo Vocational Monitoring Survey (BVMS). BVMS includes four sections: [a] demographics and disease characteristics, [b] self-reported symptom inventories, [c] general employment information, and [d] work-related problems/accommodations. Vocational status (employed vs. unemployed) will be taken from this survey.
Time Frame: 0, 12, and 24 months
Population: Patient discontinuations, withdrawals, and loss-to-follow-ups account for declining numbers in each group as study progressed.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsing MS Patients | Healthy Controls
Number analyzed (Participants) | 30 | 30
Participants
  Month 0: Employed | 14 | 30
  Month 0: Unemployed | 16 | 0
  Month 12: number analyzed (Participants) | 16 | 23
  Month 12: Employed | 7 | 21
  Month 12: Unemployed | 9 | 2
  Month 24: number analyzed (Participants) | 8 | 17
  Month 24: Employed | 3 | 16
  Month 24: Unemployed | 5 | 1

ADVERSE EVENTS:
Time Frame: 6 years total of study activity.
Groups:
- Healthy Controls: This sample 30 healthy control volunteers, matched on demographics with the multiple sclerosis group. This healthy control group was not prescribed Aubagio.
Arm/Group | MS Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 10/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MS Group (N=30) | Healthy Controls (N=30)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Minor Hair Loss (General disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Swelling in legs and feet (General disorders) | 3 (3) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT02651545/Prot_SAP_000.pdf